CLINICAL TRIAL: NCT02524041
Title: Association Between Serum Periostin Levels and Cortical Porosity in Patients With Secondary Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1308046; 130560B-22 (Other: ANSM)
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Hyperparathyroidism
Keywords: Hyperparathyroidism; microarchitecture; periostin
MeSH Terms: conditions — Hyperparathyroidism | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- secondary hyperparathyroidism (Experimental): Blood specimen and HR-pQCT for measure bone quality and quantity
  Interventions: Device: HR-pQCT; Other: blood specimen

INTERVENTIONS:
Device: HR-pQCT — The Xtrem CT scanco device is a HR-pQCT used for 3D bone measurements at the tibia and the radius levels in humans
  Other Names: Xtrem CT scanco
Other: blood specimen — blood specimen

SUMMARY:
Based on the evidence that periostin is specifically involved in intra-cortical remodeling control, our working hypothesis is that assessment of its concentration in the serum would be helpful in identifying patients with severe cortical porosity, a critical parameter in bone fragility. Periostin expression by osteoblasts and osteocytes is part of the bone cortical response to anabolic stimuli such as mechanical strain or intermittent increase in parathyroid hormone. However, it remains unknown whether this expression may participate as well to mechanisms that will lead to exaggerated intra-cortical remodeling and subsequent bone loss.

In rare clinical situations in which trans-iliac bone biopsies will be necessary to better understand their bone status in addition to densitometry and biological bone markers assessment, specific analyses using immune-staining techniques will be performed on the bone sample. Data from routine follow-up every six months will be also collected in this specific sub-group.

High resolution peripheral quantitative computerized tomography (HR-pQCT) gives the opportunity of performing a virtual bone biopsy providing information on trabecular and cortical microarchitecture in vivo. These microarchitectural parameters allow a more accurate evaluation of the alteration of the bone structure and therefore of the fracture risk as compared to current tools used in clinical practice such as densitometry. However, the availability of such HRpQCT facilities is limited and there is on-going development on the best way of measuring porosity for example. The definition of a biological profile including key proteins such as periostin and sclerostin involved in porosity mechanisms is therefore of great interest. A better understanding of the relationship between bone matrix components and parathyroid hormone effects also appears as critical. Follow-up of routine evaluation parameters reflecting bone status in a subgroup of specific patients could also provide new and additional information.

ELIGIBILITY:
Inclusion Criteria:

* Hyperparathyroidism defined by a parathyroid hormone serum level above 65 ng/ml, secondary to Chronic Kidney Disease (CKD) ou vitamin D deficiency

Exclusion Criteria:

* Concurrent bone disease (such as Paget's disease, osteomalacia),
* Other endocrinopathy having an impact on bone metabolism (such as Cushing, hyperthyroidism, severe hypogonadism (except menopause)),
* Current or previous bisphosphonate treatment.
* Transplantation
* parathyroidectomy
* Life expectancy less than 3 months.
* Lack of study understanding.
* Lack of agreement.
* Under legal control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Correlation between periostin level and cortical porosity | day 1
  Correlation between periostin serum level (ng/ml) and cortical porosity. Cortical porosity (%) is measured by HR-pQCT

SECONDARY OUTCOMES:
Correlation between periostin level and other trabecular and cortical microarchitectural parameters (composite outcome) | day 1
  Correlation between periostin serum level (ng/ml) and other trabecular and cortical microarchitectural parameters. Cortical microarchitectural parameters are a composite measure measured by HR-pQCT. The measures are : Total volumetric mineral density (mg/ccm HA), Trabecular volumetric mineral density (mg/ccm HA), Cortical volumetric mineral density (mg/ccm HA), Number of bone trabeculae (1/mm), Trabecular thickness (mm), Cortical thickness (mm), Trabecular spacing (mm)
  o Trabecular distribution (mm)
Correlation between parathyroid hormon level and other trabecular and cortical microarchitectural parameters (composite outcome) | day 1
  Correlation between parathyroid hormon serum level (pg/ml) and other trabecular and cortical microarchitectural parameters. Cortical microarchitectural parameters are a composite measure measured by HR-pQCT. The measures are : Total volumetric mineral density (mg/ccm HA), Trabecular volumetric mineral density (mg/ccm HA), Cortical volumetric mineral density (mg/ccm HA), Number of bone trabeculae (1/mm), Trabecular thickness (mm), Cortical thickness (mm), Trabecular spacing (mm)
  o Trabecular distribution (mm)
Correlation between Sclerostin serum level and cortical porosity | Day 1
  Correlation between Sclerostin serum level (ng/ml) and cortical porosity.Cortical porosity (%) is measured by HR-pQCT.
Correlation between parathyroid hormon level and cortical porosity | Day 1
  Correlation between parathyroid hormon serum level (pg/ml) and cortical porosity.Cortical porosity (%) is measured by HR-pQCT.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THOMAS, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France